CLINICAL TRIAL: NCT00780182
Title: An Open-Label, Randomized, 3-Way Crossover, Single-Dose Study in Healthy Volunteers Comparing the Bioavailability of CMX001 (HDP-Cidofovir Conjugate) Delivered as a Tablet Formulation vs a Solution Formulation and the Effect of Food on CMX001 Bioavailability
Brief Title: Comparative Bioavailability and Effect of Food on CMX001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Neil Frazer/ Chief Medical Officer, Chimerix
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CMX001-103; DMID-08-0020
Record Dates: First submitted 2008-10-23; First posted 2008-10-27 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Bioavailability
MeSH Terms: interventions — brincidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All subjects will receive three 40mg doses of CMX001 as 1)solution fasted, 2)tablet fasted and 3)tablet following a high-fat breakfast. The order in which each subject receives each of the doses will be determined by a randomization code.
  Interventions: Drug: CMX001

INTERVENTIONS:
Drug: CMX001 — CMX001 tablet fasted, CMX001 tablet fed, CMX001 solution fasted

SUMMARY:
The purpose of this study is to compare the bioavailability of CMX001 when administered as a tablet vs a solution and to determine the effect of a high-fat meal on CMX001 bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-childbearing females 18-55 years old

Exclusion Criteria:

* Use of an investigational drug and/or treatment within 30 days prior to enrollment.
* Positive HIV, Hepatitis B or Hepatitis C test result
* Tobacco user
* History of GI disease or disorder
* History of positive fecal occult blood test (FOBT)
* Body Mass Index (BMI) > 30 or < 18, or body weight < 50 kg
* Prior abdominal or pelvic surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
AUC and Cmax of CMX001 and cidofovir | Each of 3 doses

SECONDARY OUTCOMES:
Clinical and laboratory endpoints and adverse events | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Evin H Sides, III, MD, Principal Investigator — AAIPharma
Locations (1):
- AAI Pharma, Rtp, North Carolina, United States